CLINICAL TRIAL: NCT01082471
Title: A Randomised Double-blind Study to Compare the Analgesic Efficacy and Safety Profiles of M6G and Morphine, as a Loading Dose Followed by PCA, in Patients Suffering Moderate to Severe Post-operative Pain Requiring PCA for at Least 24 Hours
Brief Title: An Efficacy and Safety Study to Compare Morphine 6-glucuronide (M6G) and Morphine in Patients Suffering With Post-Operative Pain for at Least 24 Hours
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Paion UK Ltd. (Industry)
Collaborators: Chiltern International Ltd. (Industry); HFL Ltd. (Unknown)
Responsible Party: Dr. Alexander Binning, Western Infirmary, Glasgow, NHS Scotland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M6G022; 2005-001690-99 (EudraCT Number)
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Pain
Keywords: Morphine 6-glucuronide; Morphine; Patient Controlled Analgesia; Post Operative Nausea and Vomiting
MeSH Terms: conditions — Pain, Postoperative; Vomiting | interventions — morphine-6-glucuronide; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- M6G (Experimental): An initial slow bolus injection up to 60 min prior to end of surgery. If required, two additional slow bolus injections to achieve baseline pain relief. Continuing on PCA for a minimum of 24 hours.
  Interventions: Drug: Morphine 6-glucuronide
- Morphine (Active Comparator): An initial slow bolus injection up to 60 min prior to end of surgery. If required, two additional slow bolus injections to achieve baseline pain relief. Continuing on PCA for a minimum of 24 hours.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Morphine 6-glucuronide
  Arms: M6G
Drug: Morphine
  Arms: Morphine

SUMMARY:
To compare the incidence and severity of nausea in the study treatment groups, during the 18-hour period starting 6 hours after titration to pain relief; following confirmation of the assumption of non-inferiority between the two groups of pain relief over the 24 hour post-operative period. Pain relief and nausea will be determined by measuring the areas under the curves of pain intensity and nausea verbal rating scale scores.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients undergoing any of the following elective surgical procedures that, in the Investigator's opinion, would have required the use of post-operative patient controlled analgesia for a minimum of 24 hours:
* Abdominal hysterectomy with the exception of laparoscopic procedures.
* Bowel / gastrointestinal (GI) surgery
* Major urological surgery
* Aged ≥ 18 years
* American Society of Anesthesiologists (ASA) grades I to III
* If female, the patient had to be post-menopausal (last menstruation > 1 year previously), or surgically sterile (e.g. full hysterectomy or tubal ligation). If neither of these was the case, she had to use adequate contraception (i.e. hormonal contraceptive, intrauterine device (IUD), or a double barrier method) and to have a negative urine pregnancy test during the 24-hours prior to surgery.
* Provide written informed consent to participate in the trial prior to surgery.

Exclusion Criteria:

* The patient was pregnant or lactating.
* Had a known sensitivity to morphine or other opiates, or a medical condition such that opiates were contraindicated.
* Had a known sensitivity to paracetamol, or a medical condition such that paracetamol was contraindicated.
* Had received any investigational drug within the 90 days prior to the start of the study, or was scheduled to receive one during the study period.
* Had been involved in any previous M6G study.
* Had a documented history or current evidence of alcohol or drug abuse within the year prior to screening.
* Had clinically significant findings on pre-treatment evaluations (e.g. laboratory results, electrocardiograms, medical history, physical examination) that, in the Investigator's opinion, should have excluded them from the study.
* Had a concurrent disorder that resulted in excessive pain that, in the Investigator's opinion, would have interfered with the pain assessments during the study (e.g.severe rheumatoid arthritis, muscle dystrophy or neuropathic pain).
* Had a blood clotting disorder or other blood dyscrasias.
* Had requested the use of epidural or intrathecal anaesthesia techniques.
* Required the use of a local anaesthetic block and/or infiltration of wound sites.
* Required the concomitant use of opioids or non-steroidal anti-inflammatory drugs(NSAIDs) during the study due to an existing concurrent condition.
* Had a history of Left Ventricular Failure or compromised cardiovascular function, defined as New York Heart Association (NYHA) level 3.
* Had a history of severe renal impairment or a creatinine level > 3 times the upper limit of normal.
* Was having surgery that would have prevented the use of oral or rectal paracetamol(iv administration of paracetamol was not allowed).
* Was expected to require prolonged ventilation after surgery.
* Was opioid tolerant or had a history of chronic opioid use.
* Had cognitive impairment that would, in the Investigator's opinion, have precluded participation or compliance with protocol defined procedures (i.e. use of PCA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 517 (Actual)
Dates: Start 2005-11; Primary Completion 2006-11 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of nausea | The 6-18 hour period after titration to pain relief
  To compare the incidence and severity of nausea in the study treatment groups, during the 18-hour period starting 6 hours after titration to pain relief; following confirmation of the assumption of non-inferiority between the two groups of pain relief over the 24-hour post-operative period. Pain relief and nausea were determined by measuring the areas under the curves of pain intensity and nausea verbal rating scale scores.

SECONDARY OUTCOMES:
Analgesic effect | 0-48 hours after titration to pain relief
  To compare the analgesic effect of the study treatments using an Investigator- and patient-administered VRS-11 scale of pain intensity over the following time periods following achievement of baseline pain relief.
  1. 0-12 hours (AUCbaseline-12)
  2. 0-48 hours (AUCbaseline - 48)
  3. 12-24 hours (AUC12 - 24)
  4. 24-48 hours (AUC24 - 48) Pain levels will be compared using the AUC from baseline.
The incidence and severity of nausea | 0-48 hours
  To compare the incidence and severity of nausea in the study treatment groups over the following time periods following achievement of baseline pain relief: 0-12 hours, 0-24 hours, 0-48 hours, 12-24 hours, 24-48 hours.
The incidence and severity of vomiting | 0-48 hours
  To compare the incidence and severity of vomiting in the study treatment groups over the following time periods following achievement of baseline pain relief: 0-12 hours, 0-24 hours, 0-48 hours, 12-24 hours, 24-48 hours
The amounts of study drug required to achieve a baseline pain severity score of ≤ 3 | 60-30mins before close of surgery to time 0.
  To compare the amounts of study drug required to achieve a baseline pain severity score of ≤ 3

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Binning, M.D., Principal Investigator — Intensive Care Unit, Level 5, Western Infirmary, Glasgow, G11 6NT; James Lees, B.Sc., Study Director — Paion UK Ltd.
Locations (7):
- Teaching Hospital Bulovka, Department of Urology, Prague, Czechia
- Anaesthetisia - Resuscitation Department, Tenon Hospital, Paris, Cedex 20, France
- Universitätsklinikum Bonn, Klinik und Poliklinik f. Anaesthesiologie, Bonn, Germany
- Department of Anaesthesiology, Leiden University Medical Centre, Leiden, Netherlands
- Ii Klinika Anestezjologii i It, Lublin, Poland
- United Kingdom (2):
  - Intensive Care Unit, Level 5, Western Infirmary,, Glasgow, Renfrewshire
  - St John's Hospital, Livingston, West Lothian